CLINICAL TRIAL: NCT02577016
Title: A Phase III, Multicenter, Randomized, Placebo-Controlled, Parallel-Group, Double-Blind Trial to Assess the Safety and Efficacy of Addition of Sitagliptin in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Ipragliflozin Monotherapy in Addition to Diet and Exercise Therapy
Brief Title: Double-blind Sitagliptin Add-on Study in Japanese Participants With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Ipragliflozin (MK-0431J-842)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431J-842; 153096 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2015-10-14; First posted 2015-10-15 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin + Ipragliflozin (Experimental): Sitagliptin, oral, once daily for 24 weeks plus ipragliflozin (base therapy), in addition to diet and exercise.
  Interventions: Drug: Sitagliptin; Drug: Ipragliflozin
- Placebo + Ipragliflozin (Active Comparator): Placebo to sitagliptin, oral, once daily for 24 weeks plus ipragliflozin (base therapy), in addition to diet and exercise.
  Interventions: Drug: Placebo; Drug: Ipragliflozin

INTERVENTIONS:
Drug: Sitagliptin — 50 mg tablet administered orally
  Other Names: Januvia®, Tesavel®, Xelevia®, Ristaben®, Glactiv®
  Arms: Sitagliptin + Ipragliflozin
Drug: Placebo — Placebo to sitagliptin administered orally
  Arms: Placebo + Ipragliflozin
Drug: Ipragliflozin — 50 mg tablet administered orally as background medication

SUMMARY:
This is a study to assess the safety and efficacy of the addition of sitagliptin in Japanese participants with Type 2 diabetes mellitus (T2DM) who have inadequate glycemic control on ipragliflozin, diet, and exercise therapy. The primary hypothesis of the study is that the addition of sitagliptin once daily compared with placebo provides greater reduction in hemoglobin A1C (HbA1c) as assessed by change from baseline (Week 0) to Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Inadequate glycemic control on diet/exercise therapy and ipragliflozin monotherapy
* HbA1c ≥7.0% and ≤10.0% before study start

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of any of the following medications: thiazolidinediones (TZD) and/or insulin within 12 weeks prior to study participation, sitagliptin within 8 weeks prior to study participation.
* Currently has a urinary tract infection or genital infection with subjective symptom

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Seino Y, Kaku K, Kadowaki T, Okamoto T, Sato A, Shirakawa M, O'Neill EA, Engel SS, Kaufman KD. A randomized, placebo-controlled trial to assess the efficacy and safety of sitagliptin in Japanese patients with type 2 diabetes and inadequate glycaemic control on ipragliflozin. Diabetes Obes Metab. 2021 Jun;23(6):1342-1350. doi: 10.1111/dom.14346. Epub 2021 Feb 28. PMID 33565686

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, all participants received placebo for 2 weeks.
Period: Overall Study
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Started | 70 | 71
Completed | 68 | 69
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin | Total
Number analyzed (Participants) | 70 | 71 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (11.6) | 54.0 (9.5) | 55.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 54 | 45 | 99
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.01 (0.81) | 8.08 (0.79) | 8.04 (0.80)
2-hour postmeal glucose (2-hr PMG) [Mean (Standard Deviation); unit: mg/dL] — Population: All randomized participants with baseline 2-hr PMG measurement.
  mg/dL
    number analyzed (Participants) | 70 | 70 | 140
    (all) | 211.9 (49.8) | 215.3 (47.0) | 213.6 (48.3)
Glucose total AUC0-2hr after meal [Mean (Standard Deviation); unit: mg･hr/dL] — Population: All randomized participants with baseline Glucose total AUC0-2hr after meal measurement.
  mg･hr/dL
    number analyzed (Participants) | 70 | 70 | 140
    (all) | 414.4 (73.8) | 422.5 (68.2) | 418.5 (70.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: md/dL] | 148.8 (25.4) | 151.2 (27.0) | 150.0 (26.1)
Prior use of other antihyperglycemic agents (AHAs) [Count of Participants; unit: Participants] — Other AHAs refers to the use of AHAs other than sodium-glucose cotransporter 2 (SGLT2) inhibitors within 8 weeks of study start.
  Participants
    Yes | 24 | 25 | 49
    No | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c at Week 24
Description: HbA1c is measured as percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent. Statistical analysis based on a constrained longitudinal data analysis (cLDA) model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, and treatment by time by prior use of AHAs with the constraint that the mean baseline is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of HbA1c (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Number analyzed (Participants) | 70 | 71
Percent | -0.69 [-0.85 to -0.53] | 0.14 [-0.02 to 0.29]
Statistical Analysis 1: Comparison: Sitagliptin + Ipragliflozin vs Placebo + Ipragliflozin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -0.83, 95% CI 2-sided [-1.05 to -0.62]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 26 weeks
Population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Number analyzed (Participants) | 70 | 71
Percentage of participants | 54.3 | 63.4

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Number analyzed (Participants) | 70 | 71
Percentage of participants | 2.9 | 0.0

4. Secondary Outcome: Change From Baseline in 2-hr PMG at Week 24
Description: Change from baseline in 2-hr PMG at Week 24 is defined as Week 24 2-hr PMG minus Week 0 2-hr PMG. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, and treatment by time by prior use of AHAs with the constraint that the mean baseline 2-hr PMG is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of 2-hr PMG (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Number analyzed (Participants) | 70 | 71
mg/dL | -39.0 [-48.1 to -29.9] | 3.4 [-5.5 to 12.3]
Statistical Analysis 1: Comparison: Sitagliptin + Ipragliflozin vs Placebo + Ipragliflozin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -42.5, 95% CI 2-sided [-53.7 to -31.2]

5. Secondary Outcome: Change From Baseline in Glucose Total Area Under the Plasma Concentration Curve From Hour 0 to Hour 2 (AUC0-2hr) After Meal at Week 24
Description: Change from Baseline in Glucose Total AUC0-2hr after Meal at Week 24 is defined as Week 24 Glucose Total AUC0-2hr after a meal minus Week 0 Glucose Total AUC0-2hr after a meal. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, and treatment by time by prior use of AHAs with the constraint that the mean baseline glucose total AUC0-2hr after meal is the same for both treatment groups.
Time Frame: Baseline and Week 24 (just before loading meal [0 min], 30 min, 60 min and 120 min)
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of glucose total AUC0-2hr after meal (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg･hr/dL
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Number analyzed (Participants) | 70 | 71
mg･hr/dL | -65.7 [-79.2 to -52.2] | 1.3 [-11.9 to 14.5]
Statistical Analysis 1: Comparison: Sitagliptin + Ipragliflozin vs Placebo + Ipragliflozin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -67.0, 95% CI 2-sided [-84.0 to -50.0]

6. Secondary Outcome: Change From Baseline in FPG at Week 24
Description: Change from baseline in FPG at Week 24 is defined as Week 24 FPG minus Week 0 FPG. Statistical analysis based on a cLDA model with terms for treatment, time, prior use of AHAs, the interactions of treatment by time, time by prior use of AHAs, and treatment by time by prior use of AHAs with the constraint that the mean baseline FPG is the same for both treatment groups.
Time Frame: Baseline and Week 24
Population: All randomized participants who received at least one dose of treatment period study medication and have at least one measurement of FPG (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Number analyzed (Participants) | 70 | 71
mg/dL | -11.8 [-16.3 to -7.4] | -0.6 [-5.0 to 3.8]
Statistical Analysis 1: Comparison: Sitagliptin + Ipragliflozin vs Placebo + Ipragliflozin; Test type: Superiority; p < 0.001, Constrained longitudinal data analysis; Based on a cLDA model with the terms listed above; Difference in least squares means = -11.2, 95% CI 2-sided [-17.2 to -5.2]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | Sitagliptin + Ipragliflozin | Placebo + Ipragliflozin
Serious Adverse Events (participants affected / at risk) | 3/70 | 0/71
Other Adverse Events (participants affected / at risk) | 10/70 | 18/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin + Ipragliflozin (N=70) | Placebo + Ipragliflozin (N=71)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin + Ipragliflozin (N=70) | Placebo + Ipragliflozin (N=71)
Nasopharyngitis (Infections and infestations) | 6 (7) | 18 (24)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.